CLINICAL TRIAL: NCT06519773
Title: Modified Periosteal Inhibition Utilizing Bone Graft Versus Collagen Sponge with Simultaneous Implant Placement in Aesthetic Zone
Brief Title: Modified Periosteal Inhibition with Simultaneous Implant Placement in Aesthetic Zone
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ghadeer Khalil Elbagoory, Associate lecturer, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OMPDR 4-24 2191
Record Dates: First submitted 2024-07-16; First posted 2024-07-25 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Immediate Dental Implant
Keywords: Immediate implant; Modified periosteal inhibition

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Twenty surgical sites will be divided into two groups; each of which has ten surgical sites. Grouping will be done randomly sequentially numbered, opaque, sealed envelopes (SNOSE)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Collagen sponge group : (Sham Comparator): ten sites will be treated by MPI technique+ cortical lamina membrane and collagen sponge.
  The jumping gap between implant and buccal plate of bone will be filled with collagen sponge.
  Interventions: Procedure: Modified periosteal inhibition
- Bone graft group: (Active Comparator): ten sites will be treated by MPI technique +cortical lamina membrane and xenograft collagen.
  The jumping gap between implant and buccal plate of bone will be filled with xenograft collagen.
  Interventions: Procedure: Modified periosteal inhibition

INTERVENTIONS:
Procedure: Modified periosteal inhibition — After local anathesia, a traumatic extraction of the hopeless tooth will be made trying as much as possible to preserve the labial plate of bone and overlying soft tissue.
  * Once the tooth is extracted, the socket is gently debrided and irrigated using sterile saline solution. Then the dental implant is placed in the best prosthetic driven position, following the guidelines for immediate implants using prefabricated computer guided surgical template.
  * After accurate implant placement, a full-thickness flap will be elevated at mesial and distal papilla making a buccal envelope. A soft bone lamina will be trimmed and hydrated in sterile saline solution for 30 s to soften it; it should be 1-2 mm larger and deeper than the vestibular bone. Then the jumping gap between the dental implant and the buccal plate of bone will be filled using either collagen sponge or xenograft.

SUMMARY:
A randomized controlled clinical and radiographic trial. Twenty sites with remaining roots or non-restorable teeth in the maxillary anterior region that fulfill the inclusion criteria will be selected from the Periodontology Clinic, Faculty of Dentistry, Tanta University. These sites will be divided into two groups; each of which has ten surgical sites. After phase I therapy, a traumatic extraction of the hopeless tooth will be made trying as much as possible to preserve the labial plate of bone and overlying soft tissue.

* Once the tooth is extracted, the socket is gently debrided and irrigated using sterile saline solution. Then the dental implant is placed in the best prosthetic driven position, following the guidelines for immediate implants using prefabricated computer guided surgical template.
* After accurate implant placement, a full-thickness flap will be elevated at mesial and distal papilla making a buccal envelope. A bone lamina 0.5 mm thickness will be trimmed and hydrated in sterile saline solution for 30 s to soften it; it should be 1-2 mm larger and deeper than the vestibular bone.

DETAILED DESCRIPTION:
A randomized controlled clinical and radiographic trial. The purpose of the present study will be explained to the patients and informed consents will be obtained according to guidelines adopted by the Research Ethics Committee, Faculty of Dentistry, Tanta University. Twenty sites with remaining roots or non-restorable teeth in the maxillary anterior region that fulfill the inclusion criteria will be selected from the Periodontology Clinic, Faculty of Dentistry, Tanta University. Twenty surgical sites will be divided into two groups; each of which has ten surgical sites. Grouping will be done randomly sequentially numbered, opaque, sealed envelopes (SNOSE).

1. Phase I therapy

   * Full mouth supra and subgingival scaling and root planing will be performed to all enrolled patients. Patients will be instructed to rinse twice daily with 0.12% chlorohexidine mouth wash for 2 weeks.
   * Before tooth extraction, initial radiographic records by cone beam computed tomography (CBCT) scans of the maxillary arch will be made. The pre-extraction measurements will be taken from CBCT scans to evaluate the presence of a fully intact labial plate of bone ≤1 mm. The labial plate thickness of the tooth to be extracted will be measured on cross sectional cuts at three levels below the labial bone crest: 0, 2, and 5 mm.
2. Surgical technique:

   * After local anathesia, a traumatic extraction of the hopeless tooth will be made trying as much as possible to preserve the labial plate of bone and overlying soft tissue.
   * Once the tooth is extracted, the socket is gently debrided and irrigated using sterile saline solution. Then the dental implant provided by Bego Dental Implant is placed in the best prosthetic driven position, following the guidelines for immediate implants using prefabricated computer guided surgical template.
   * After accurate implant placement, a full-thickness flap will be elevated at mesial and distal papilla making a buccal envelope. A soft bone lamina provided by osteobiol 0.5 mm thickness will be trimmed and hydrated in sterile saline solution for 30 s to soften it; it should be 1-2 mm larger and deeper than the vestibular bone. The cortical lamina will be fixed using Glubran 2 provided by GEM which is N-butyl 2 cyanoacrylate + Metacryloxysulfolane adhesive.

   The labial gap will be filled either with bone graft ( Regeinoss cortico cancelleous granules with collagen- xenograft. GRANNTIE )or collagen sponge.

   The socket orifice will be sealed using a customized healing abutment screwed to the implant, adequately finished, and polished to ensure a proper soft tissue emergence profile. The papilla will be sutured back using 5.0 polypropylene sling suture. For all cases, the sutures will be removed after 2 weeks.
3. Postoperative Phase -All subjects will receive postoperative instructions including:

   * Rinsing with 0.1% Chlorhexidine mouth rinse twice daily for two weeks.
   * Antibiotics combination of 500 mg Metronidazole along with Amoxicillin Clavulanate (Augmentin 1g) every 12 hours one day preoperatively and continuing for 5 days after extraction.
   * Non-steroidal anti-inflammatory (NSAID) medication of Ibuprofen 400 mg twice daily for one week.

ELIGIBILITY:
Inclusion Criteria:

1. Intact labial plate of bone with thickness ≤1 mm (Socket type I).
2. Moderate to thick gingival phenotype.
3. Bone quality ranges from D2-D3 as gained from preoperative cone beam computed tomography.
4. Presence of at least 3 mm of keratinized gingiva.
5. Optimal compliance as evidenced by no missing treatment appointments and positive attitude towards oral hygiene.

Exclusion Criteria:

1. Medically compromised patients and systemic conditions precluding implant and periodontal surgery.
2. Pregnant or lactating women.
3. Smoking
4. Absence of buccal plate of bone.
5. History of chemotherapy, radiotherapy in head and/or neck region.
6. Bisphosphonate therapy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Radiographic cone beam computed tomography (CBCT) assessment | baseline, 6 and 12 months after implant placement.
  The primary outcome of the study is to assess the amount of bone formed labial to the implant on the CBCT. This will be made by measuring bone thickness at the bone crest, 2mm and 5 mm above the crest

SECONDARY OUTCOMES:
Implant stability | baseline and 6 months after implant placement.
  The implant stability: it will be measured using the Resonance Frequency Analysis Device.
Soft tissue healing | within one week after surgery, 1 month and 6 months
  it will be recorded according to soft tissue healing index Score Clinical finding Very poor • Tissue colour: ≥50% of gingiva red
  * Response to palpation: Bleeding.
  * Granulation tissue: Present
  * Incision margin: Not epithelialized, with loss of epithelium beyond incision margin.
  * Suppuration: Present. Poor • Tissue colour: ≥50% of gingiva red.
  * Response to palpation: Bleeding.
  * Granulation tissue: Present.
  * Incision margin: Not epithelialized, with connective tissue exposed Good • Tissue colour: ≥25% and<50% of gingiva red
  * Response to palpation: No bleeding.
  * Granulation tissue: None
  * Incision margin: No connective tissue exposed. Very good • Tissue colour: <25% of gingiva red.
  * Response to palpation: No bleeding.
  * Granulation tissue: None
  * Incision margin: No connective tissue exposed. Excellent • Tissue colour: All tissues pink.
  * Response to palpation: No bleeding.
  * Granulation tissue: None
  * Incision margin: No connective tissue exposed.
The esthetic | immediately after final prosthetic delivery and 6 months later.
  it will be evaluated by pink esthetic score (PES) Variables 0 1 2 Mesial papilla Shape vs. reference tooth Absent Incomplete Complete Distal papilla Shape vs. reference tooth Absent Incomplete Complete Level of soft-tissue margin Level vs. reference tooth Major discrepancy > 2mm Minor discrepancy 1-2 mm No discrepancy < 1mm Soft-tissue contour Natural, matching reference tooth Unnatural Fairly natural Natural Alveolar process Alveolar process deficiency Obvious Slight None Soft-tissue color Color vs. reference tooth Obvious difference Moderate difference No difference Soft-tissue texture Texture vs. reference tooth Obvious difference Moderate difference No difference
  * Each variable will take a score from: 2-1-0, with 2 being the best and 0 being the poorest score.
  * The highest possible score reflecting a perfect match of the peri-implant soft tissue with that of the reference tooth is 14 for all the seven parameters.
Digital Assessment | baseline, 6 and 12 months.
  Each group will be subjected to intraoral scanning at baseline, 6 and 12 months. After loading The changes in peri-implant mucosal level will be assessed by superimposition of scanning files of different intervals to monitor the vertical and horizontal linear measurement of the mucosa calculated by software.

CONTACTS AND LOCATIONS:
Overall Officials: Ghadeer Elbagoory, Msc, Study Chair — Tanta University
Locations (1):
- ElGharbiya, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No